CLINICAL TRIAL: NCT05534854
Title: Frequency, Clinical Phenotype and Genetic Analysis of Heritable Kidney Cancer Syndromes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Zhejiang Provincial People's Hospital (Other); Tongji Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai 10th People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RENJI-IKCS
Record Dates: First submitted 2022-07-04; First posted 2022-09-10 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Renal Tumor Histology; Kidney Cancer; Renal Cell Carcinoma; Familial Renal Cancer; HLRCC; VHL Syndrome; BAP1 Tumor Predisposition Syndrome; FLCN Gene Mutation; ALK Gene Mutation; FH Gene Mutation; Birt-Hogg-Dube Syndrome; MET Gene Mutation; Cutaneous Leiomyoma; Cutaneous Leiomyomata With Uterine Leiomyomata
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; von Hippel-Lindau Disease; Birt-Hogg-Dube Syndrome; Hereditary leiomyomatosis and renal cell cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with heritable kidney cancer syndrome: Patients with known or suspected heritable kidney cancer syndromes, including VHL and HLRCC Disease.
  Interventions: Genetic: Gene test
- Family members of heritable kidney cancer syndrome: Family members (related by blood) of patients who have or are suspected of having heritable kidney cancer syndromes, including VHL and HLRCC Disease.
  Interventions: Genetic: Gene test
- Not proven genetic etiology: Patients and biologic family members with a heritable kidney cancer syndrome of suspected, but not proven genetic etiology.
  Interventions: Genetic: Gene test

INTERVENTIONS:
Genetic: Gene test — Next generation sequencing of blood, urine and/or benign and malignant tissue of patients and family members with known or suspected heritable kidney cancer syndromes, including VHL and HLRCC Disease.

SUMMARY:
This study will investigate the frequency, clinical phenotype, management and molecular genetic defects of heritable kidney cancer syndromes. Families with kidney cancer with known or suspected genetic basis will be enrolled. Affected individuals or individuals suspected of having a germline kidney cancer will undergo periodic clinical assessment and genetic analyses for the purpose of: 1) definition and characterization of phenotype, 2) determination of the natural history of the disorder, and 3) genotype/phenotype correlation. Genetic linkage studies may be performed in situations in which the genetic basis of the disorder has not been elucidated. This research will have a significant impact on the overall management of heritable kidney cancer syndromes patients and family members who are at risk for heritable kidney cancer syndromes. The study will ultimately facilitate the development of novel screening, prevention and treatment strategies for these individuals with the syndrome. In addition this study could have impact on the management of patients with personal and/or family history of heritable kidney cancer syndromes.

DETAILED DESCRIPTION:
Background:

• The genetic etiology of heritable kidney cancer syndromes remains to be determined.

Objectives:

* Define the risk of developing renal cance in heritable kidney cancer syndromes
* Define the types and characteristics (including patterns of growth) of heritable kidney cancer syndromes.
* Determine genotype/phenotype correlations.
* To characterize the natural and clinical histories of heritable kidney cancer syndromes.
* To determine the genetic etiology of heritable kidney cancer syndromes.

Design:

* These rare families will be recruited to genetically confirm diagnosis, determine size and location of renal tumors, size at presentation, growth rate and metastatic potential of renal tumors.
* Genetic testing will be offered to gain appreciation of the effect of mutations on the relative activity of various germline and somatic mutations.
* To determine if there is a relationship between mutation and disease manifestations and phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to 2 years of age. All patients and guardians (for children younger than 18 years of age) must sign an informed consent document indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed. Patients under the age of 18 but who are age 13 or older will be asked to sign an assent document prior to participation.
* Individuals and biologic family members with a suspected or an established diagnosis of a heritable kidney cancer syndrome in which the disease gene is known, including von Hippel-Lindau (VHL) and hereditary papillary renal carcinoma (HPRC).
* Individuals and biologic family members with a suspected or an established diagnosis of a heritable kidney cancer syndrome in which the disease gene is not yet known, specifically hereditary forms of Type II papillary renal cancer, clear cell renal carcinoma, renal oncocytoma, chromophobe renal carcinoma or Birt Hogg Dube.
* Individuals and biologic family members who have heritable kidney cancer syndromes of suspected, but not proven genetic etiology, including families with more than one individual affected by the same or related cancers.
* Subject Enrollment Categories (to include both affected and unaffected biologic relatives).

Exclusion Criteria:

* Pregnant women are excluded from enrollment onto this study because there is no direct benefit for participating in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected heritable kidney cancer syndromes and their biologic family members with heritable kidney cancer syndromes will be recruited primarily from the urology, oncology, and genetics communities worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotypes of patients of heritable kidney cancer syndromes | 5 years
  Chart review of disease outcome
Genotypes of patients of heritable kidney cancer syndromes | 5 years
  Genotyping for genetic variants that could modify the risk of cancer in subjects.

SECONDARY OUTCOMES:
Clinical phenotypes of family members of the patients | 5 years
  Questionnaire and chart review of the clinical phenotype
Prevalence of germline variants in the unselected general population of renal cancer patients | 5 years
  Frequency of germline pathogenic/likely pathogenic variants in renal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Study Chair — RenJi Hospital
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided